CLINICAL TRIAL: NCT06286618
Title: Moving to Integrated and Holistic Disease Prevention Among Underserved Mississippians
Brief Title: Nutrition360: Moving to Integrated and Holistic Disease Prevention Among Underserved Mississippians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Mississippi (Other)
Collaborators: My Brother's Keeper, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: HHSN268201800015I
Record Dates: First submitted 2024-02-13; First posted 2024-02-29 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-06

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychosocial or Structural Intervention (Experimental): During optimization 1 phase, participants are assigned to two groups: Psychosocial or Structural Intervention. One group will receive psychosocial support for diet only and the other will receive structural support for diet only. Each group will have three modalities.
  Interventions: Behavioral: Psychosocial Intervention; Other: Structural Intervention
- Combined Psychosocial and Structural Intervention (Experimental): The optimization 2 phase will be used to test a combined psychosocial and structural intervention, based on the most feasible selections from optimization 1 phase.During optimization 2 phase, participants will be assigned to two groups. One group will receive referral based delivery model for a combined psychosocial and structural intervention and the other group will receive an integrated delivery model for a combined psychosocial and structural intervention.
  Interventions: Other: Traditional Psychosocial+Structural; Other: Integrated Psychosocial+Structural

INTERVENTIONS:
Behavioral: Psychosocial Intervention — Psychosocial intervention is an intensive behavioral therapy intervention to address dietary behaviors. Each intervention session is a one-on-one interaction that focuses on setting individualized dietary goals and following up on them and is delivered by trained personnel. Sessions are delivered in 3 modalities which include face-to-face, phone call, and telehealth delivery. Each participant is randomly assigned to receive 4 weeks of each modality in one of the following orders: 1) Face-to-face; Telehealth; Phone Call 2) Telehealth; Phone Call; Face-to-face 3) Phone call; Face-to-face; Telehealth.
  Arms: Psychosocial or Structural Intervention
Other: Structural Intervention — The structural intervention is designed to supplement the diet with food resources via three modalities: voucher-based or F/V prescription, home meal delivery, or food bank box program. The voucher-based model includes a weekly $50 gift card with a prescription for having to eat more fruits and vegetables. The home meal delivery model includes a meal subscription that supplements the diet with two meals for two people each week (four total servings worth $65 including shipping). The food bank box program consists of participants picking up a box of food weekly from a food pantry located in the outpatient clinic. Each participant is randomly assigned to receive 4 weeks of each modality in one of the following orders: 1) Voucher; Meal Delivery; Food Box 2) Meal Delivery; Food Box; Voucher 3) Food Box; Voucher; Meal Delivery.
  Arms: Psychosocial or Structural Intervention
Other: Traditional Psychosocial+Structural — Participants will receive a combination of psychosocial and structural intervention, based on the most feasible selections from the preparation phase of the study. The intervention will initiate in a referral-based fashion in which participants will receive referral at enrollment visit.
  Arms: Combined Psychosocial and Structural Intervention
Other: Integrated Psychosocial+Structural — Participants will receive a combination of psychosocial and structural intervention, based on the most feasible selections from the preparation phase of the study. The intervention will initiate in an integrated fashion in which participants will receive immediate onboard at enrollment visit.
  Arms: Combined Psychosocial and Structural Intervention

SUMMARY:
The objective for the study is to implement a pilot study to establish essential components to address diet quality in healthcare settings and examine what value an integrated service model delivery has for the primary prevention of cardiometabolic diseases with an initial focus on dietary behaviors. This objective will be met by 1: Utilizing a multiphase optimization study design to select and optimize essential components to address diet behaviors and 2: Comparing an integrated and referral-based delivery model for healthcare-based strategies that address structural and psychosocial barriers to a healthy diet for racial/ethnic minority, marginalized and disadvantaged background young to middle aged adult populations in Mississippi.

DETAILED DESCRIPTION:
The study is designed based on the multiphase optimization strategy (MOST), which includes three phases to prepare or screen, optimize, and evaluate multiple components of an intervention. During first optimization phase, study team will conduct essential component selection by pilot testing three common strategies used in healthcare settings to deliver structural and psychosocial interventions that address diet behaviors. The second optimization phase will include pilot testing to examine the optimization of delivery mode for the essential components identified in first phase. In each phase, participants between 25 to 50 years of age who are at risk for CVD-related premature mortality will be recruited to complete a 3-month intervention in a community based clinical setting in Mississippi. The proposed project will provide foundational knowledge for components and delivery models that are the most essential and cost-effective to improve dietary behaviors among racial/ethnic minority and disadvantaged background populations in Mississippi.

ELIGIBILITY:
Inclusion Criteria:

* 25 to 50 years of age
* cardiovascular disease-related premature mortality risk (people living with HIV/AIDS or diagnosed with or familial risk for diabetes, hypertension, obesity, or Metabolic syndrome)
* internet access
* Jackson (Mississippi) metropolitan statistical area residency

Exclusion Criteria:

* cancer with active treatment
* chronic obstructive pulmonary disorder, emphysema, cystic fibrosis or any other major lung disease
* liver or kidney dysfunction, end-stage renal disease, active hepatitis,
* celiac disease, colitis, or other gastrointestinal disorders
* current pregnancy or within six months postpartum at baseline
* heavy drinking
* unintentional weight loss of more than 5% of body weight within the past six months
* recent (in the past 6 months) heart attack, stroke or other major heart surgery or event
* eating disorders (anorexia or bulimia nervosa)
* currently being treated for a fungus, bacteria, viral, or other infection due to weak immune system
* Insulin dependent diabetes

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Participant Burden | up to 12 weeks
  An existing validated tool designed to assess research participant burden (Lingler et al., 2014) for cultural and contextual appropriateness; the tool includes 21 items assessed on a 5-point Likert agreement scale and the final adapted items will be summed for a total score. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
cost effectiveness | 3 months
  Cost factors were identified by the study team during the preparation phase and measured based on personnel time, commodities, and other relevant factors for the delivery of the intervention components. Effects will then be computed based on the physical burden to determine the cost-effectiveness ratio.
session attendance | 3 months
  Participant are expected to attend 12 intervention sessions over the course of 3 months. Attendance will be recorded by the participant manager as a categorical variable (yes/no). Higher attendance will mean a better outcome.
diet quality | up to 3 months
  Dietary intake will be assessed using the NHANES Dietary Screener Questionnaire, which is a validated food frequency questionnaire assessing food intake over the past month. Participants will be asked to complete this at baseline, month 1, month 2, and post program. Increases in consumption of foods such as fruits, vegetables, whole grains, dairy/calcium and decreases in added sugars, red meat, and processed meat will mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: June Gipson, PhD, Principal Investigator — My Brother's Keeper, Inc.
Locations (1):
- The University of Southern Mississippi, Hattiesburg, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
The study is pilot in nature and is being used to support intervention development. Due to the small sample size, the data would not be suitable for secondary analysis.

REFERENCES:
- [Derived] Lemacks JL, Greer T, Aras S, Holbrook S, Gipson J. Multiphase optimization strategy to establish optimal delivery of nutrition-related services in healthcare settings: A step towards clinical trial. Contemp Clin Trials. 2024 Nov;146:107683. doi: 10.1016/j.cct.2024.107683. Epub 2024 Sep 3. PMID 39236781